CLINICAL TRIAL: NCT00609973
Title: Double-blind, Placebo Controlled, Randomized, Multicentre, Pilot Study on the Safety and Efficacy of Ciprofloxacin for Prophylactic Prevention of Postoperative Endoscopic Recurrence in Crohn's Disease Patients
Brief Title: Ciprofloxacin for the Prevention of Postoperative Endoscopic Recurrence in Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Crohn's and Colitis Foundation (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Hans Herfarth, MD, Principal Investigator, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Cipro 1.1
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-03

CONDITIONS: Crohn's Disease
Keywords: Postoperative recurrence, inflammatory bowel disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Ciprofloxacin 500 mg bid
  Interventions: Drug: Ciprofloxacin
- B (Placebo Comparator): Placebo bid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin — Ciprofloxacin 500 mg oral bid for 6 months
  Arms: A
Drug: Placebo — Placebo bid for 6 months
  Arms: B

SUMMARY:
Despite extensive medical treatment, surgical resection is required in approximately 70% of the patients at some time. However, recurrence of the disease after operation occurs in the majority of patients and is a serious limitation of surgical management. Therapeutic options to maintain postoperative clinical remission are urgently needed. Several drugs including mesalazine, antibiotics (metronidazole, ornidazole) and azathioprine or 6-mercaptopurine have been studied in the past. But the efficacy is very limited (mesalazine), overshadowed by intolerability during long-term therapy (metronidazole, ornidazole) or inconclusive (azathioprine or 6-mercaptopurine). Research demonstrating the absence of inflammation in patients with diverting ileostomy and the clinical benefit of a postoperative antibiotic therapy using metronidazole or ornidazole implicates a role of the resident bacterial flora in the postoperative relapse. Ciprofloxacin has a broad antibacterial spectrum. More interestingly it also suppresses E. coli strains, which can be found in high numbers in early and chronic ileal lesions of Crohn's disease patients Ciprofloxacin has demonstrated beneficial effects in the therapy of inflammatory bowel diseases, but the available data of the effectiveness of ciprofloxacin allow only a very limited judgement of the safety and tolerability of a 6 months therapy of ciprofloxacin. Therefore an exploratory multicenter prospective, placebo-controlled trial is planned to analyze the safety and tolerability of a 6 months therapy with ciprofloxacin compared to placebo in 40 patients (randomly assigned in a 1:1 ratio) undergoing ileocecal resection (or resection of parts of the colon). If this therapeutic regimen demonstrates tolerability, a second larger study improving the superiority of ciprofloxacin versus placebo can be initiated.

DETAILED DESCRIPTION:
Despite extensive medical treatment, surgical resection is required in approximately 70% of the patients at some time. However, recurrence of the disease after operation occurs in the majority of patients and is a serious limitation of surgical management. In this setting the bacterial flora plays an important role as demonstrated by the benefit of a postoperative antibiotic therapy with either metronidazole or ornidazole or the absence of inflammation in patients with diverting ileostomy. However, both aforementioned antibiotic regimens have numerous adverse events limiting the value of this therapy in daily clinical practice. Ciprofloxacin suppresses the gram negative aerobic bacterial flora including E.coli strains, which can be found in early and chronic ileal lesions of Crohn's disease patients. A limited number of clinical data suggest efficacy of this drug in patients with established Crohn's disease. This exploratory multicenter prospective, placebo-controlled trial will analyze the safety and tolerability of a 6 months therapy with ciprofloxacin compared to placebo in 40 patients (randomly assigned in a 1:1 ratio) undergoing ileocecal resection (or resection of parts of the colon) with primary anastomosis. No other treatments for Crohn's disease will be permitted. The primary objective of this study is to assess the safety and tolerability of a 6 months therapy of ciprofloxacin (500 mg bid) vs. placebo tablets for prevention of endoscopic recurrence in postoperative Crohn's disease patients. The secondary objectives of this study are to evaluate the endoscopic recurrence in the neoterminal ileum and at the ileocolonic anastomosis as well as the extent of colonic lesions. Additionally bioptic samples at the anastomotic site and patient DNA samples will be collected for later analysis of bacterial ribosomal 19S RNA and DNA polymorphisms (such as NOD2 or IL-23). The clinical data generated by this study will serve as a basis for a definitive clinical trial investigating the effectiveness of ciprofloxacin in the prevention of endoscopic recurrence in postoperative Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Man or woman between 18 and 70 years of age.
* Diagnosis of Crohn's disease confirmed during index surgery.
* Detailed assessment of disease localization by colonoscopy, small bowel radiography, and/or other appropriate methods (e.g., MRI, CT) within 6 months prior inclusion into the study.
* Resection for ileal or ileo-colonic Crohn's disease with ileo-colonic anastomosis (i.e., without grossly visible disease at the resection margins); neoterminal ileum should be assessable by endoscopy.
* Ability to start oral nutrition and medication intake within 14 days after index surgery.
* Negative pregnancy test at screening visit in females of childbearing potential.
* Use of appropriate contraceptive methods for females of childbearing potential and males with procreative capacity during treatment.

Exclusion Criteria:

* Short bowel syndrome.
* Previous long term therapy with ciprofloxacin (> 6 weeks prior before surgery)
* Patients in whom any visible lesions at the anastomosis were left after index surgery.
* Serious secondary illnesses of an acute or chronic nature, which in the opinion of the Investigator renders the patient unsuitable for inclusion into the study.
* Dementia
* Uncontrolled Diabetes Type I type II
* Known drug abuse
* Known parasitic disease of the digestive system
* Active replicating Hepatitis B or Hepatitis C
* HIV-infection
* Seizure disorder
* Serum creatinine levels exceeding 1.5 mg/dL or 130 μmol/L.
* Presence of an ileal or colonic stoma.
* Known previous or concurrent malignancy (other than that considered surgically cured, with no evidence for recurrence for 5 years).
* Application of non-steroidal anti-inflammatory drugs as long term treatment.
* Known intolerance/hypersensitivity to ciprofloxacin or other quinolones or drugs of similar chemical structure or pharmacological profile.
* Chronic use of CYP1A2 substrates (aminophylline, fluvoxamine, mexiletine, mirtazapine, ropinirole, tizanidine, trifluoperazine)
* Well-founded doubt about the patient's cooperation.
* Existing pregnancy, lactation, or intended pregnancy or impregnation within the next 3 months.
* Non-use of appropriate contraceptives in females of childbearing potential (e.g. condoms, intrauterine device [IUD], hormonal contraception for females, or a means of contraception for a particular patient considered adequate by the responsible investigator) during treatment.
* Participation in another clinical trial within the last 30 days, simultaneous participation in another clinical trial, or previous participation in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-05; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans H Herfarth, MD, PhD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a pilot multicenter, randomized, double-blind, placebo-controlled trial evaluating the safety and efficacy of ciprofloxacin for the prevention of postoperative recurrence in patients with CD. The study was conducted at 6 centers between January 2008 and March 2011. 33 patients were randomized.
Pre-assignment Details: There were no significants events pre-assignment
Groups:
- Cipro: Ciprofloxacin 500 mg bid
- Placebo: Placebo bid
Period: Overall Study
Arm/Group | Cipro | Placebo
Started | 17 | 16
Completed | 9 | 10
Not Completed | 8 | 6
Not completed — Adverse Event | 2 | 1
Not completed — Protocol Violation | 4 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cipro | Placebo | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Customized [Median (Full Range); unit: Years] | 33 [19 to 70] | 27 [18 to 61] | 30 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Ciprofloxacin
Description: Adverse events (AE) Discontinuation of study drug due to probably study drug related AE
Time Frame: 6 Months
Population: Intention to Treat analysis.Adverse events (AE), which were classified as probably or possibly related to the study drug.
Measure: Number; unit: Adverse events
Arm/Group | Cipro | Placebo
Number analyzed (Participants) | 17 | 16
Adverse events
  All AE | 25 | 11
  AE probably or possibly related to study drug | 9 | 1
  Participant stops study drug due to AE | 4 | 1

2. Secondary Outcome: Endoscopic Recurrence Under Postoperative Treatment With Study Medication at 6 Months
Time Frame: 6 months
Population: Endoscopy 6 months, Intention-to-Treat analysis, patients not undergoing endoscopy were assumed to have endoscopic recurrence
Measure: Number; unit: participants
Arm/Group | Cipro | Placebo
Number analyzed (Participants) | 17 | 16
participants | 11 | 11

ADVERSE EVENTS:
Arm/Group | Cipro | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/16
Other Adverse Events (participants affected / at risk) | 8/17 | 4/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cipro (N=17) | Placebo (N=16)
Anastomotic leakage (Gastrointestinal disorders) | 0 (0) | 1 (1) — Anastomotic leakage after surgery
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cipro (N=17) | Placebo (N=16)
Increase of diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Headache (General disorders) | 2 (2) | 0 (0)
Wound healing problems (General disorders) | 1 (1) | 1 (1)
Urinary tract infection (General disorders) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No